CLINICAL TRIAL: NCT02213159
Title: Intraoperative Dexmedetomidine Versus Morphine for Postoperative Analgesia After Laparoscopic Bariatric Surgery
Brief Title: Dexmedetomidine for Postoperative Analgesia After Bariatric Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANES.CZ.2
Record Dates: First submitted 2014-08-08; First posted 2014-08-11 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-01

CONDITIONS: Obesity; Sleep Apnea; Diabetes; Hypertension
Keywords: Dexmedetomidine; bariatric surgery; postoperative pain; morphine consumption; Quality of recovery
MeSH Terms: conditions — Obesity; Sleep Apnea Syndromes; Diabetes Mellitus; Hypertension; Pain, Postoperative | interventions — Dexmedetomidine; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Active Comparator): prior to anticipated end of surgery bolus of 1 microgram/kg Dexmedetomidine intravenously over 10 minutes followed by 0.5 micrograms/kilogram/hour intravenous infusion until removal of laparoscopes
  Interventions: Drug: Dexmedetomidine
- Morphine (Active Comparator): prior to anticipated completion of surgery morphine 0.08 mg/kilogram intravenous bolus over 10 minutes followed by a saline infusion until removal of the laparoscopes
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Morphine
  Arms: Morphine

SUMMARY:
The purpose of this study is to determine if Dexmedetomidine given at the end of surgery will reduce postoperative morphine consumption and improve postoperative quality of recovery as compared to morphine in patients undergoing laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
effect of Dexmedetomidine bolus on postoperative morphine requirements

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index > 40 kg/m2 or BMI > 35 kg/m2 with comorbid conditions such as hypertension, diabetes or sleep apnea
* American Society of Anesthesiologists class I or II
* Undergoing laparoscopic sleeve gastrectomy bariatric surgery

Exclusion Criteria:

* Allergy to morphine or its derivatives
* Allergy to α-2 adrenergic agonists
* weight over 180 kg
* history of uncontrolled hypertension
* heart block greater than first degree
* prolonged QT interval
* clinically significant neurologic, cardiovascular, renal, hepatic, or gastrointestinal diseases
* received an opioid analgesic medication within a 24 h period prior to surgery
* history of alcohol, drug abuse or chronic opioid intake
* history of psychiatric disorder
* pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Total dose of morphine consumed in Post Anesthesia Care Unit (PACU) | At discharge from the PACU

SECONDARY OUTCOMES:
Time to first morphine requirement in PACU | in the PACU
Numeric Rating Scale (NRS) for Pain | in the PACU and at 24 hours
NRS for nausea | in the PACU
incidence of pruritus | in the PACU
incidence of vomiting or retching | in the PACU
incidence of respiratory complications | in the PACU
time to discharge readiness in PACU | in the PACU
total morphine consumption at 24 hours | at 24 hours
Quality of Recovery (QoR-40) score at 24 hours | at 24 hours
overall satisfaction at one month | one month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carine Zeeni, M.D., Principal Investigator — AUBMC; Sahar Siddik, M.D., Principal Investigator — AUBMC
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No